CLINICAL TRIAL: NCT02092909
Title: Phase 1/2 Open-Label, Multiple-dose, Dose-escalation Study to Evaluate the Safety and Tolerability of IMO-8400 in Patients With Relapsed or Refractory Waldenstrom's Macroglobulinemia
Brief Title: Phase 1/2 Dose Escalation Study in Patients With Relapsed or Refractory Waldenstrom's Macroglobulinemia
Acronym: 8400-401
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Lack of efficacy
Sponsor: Idera Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 8400-401
Record Dates: First submitted 2014-03-18; First posted 2014-03-20 (Estimated); Results first posted 2019-08-29 (Actual); Last update posted 2019-09-10 (Actual); Status verified 2019-08

CONDITIONS: Waldenstrom's Macroglobulinemia
MeSH Terms: conditions — Waldenstrom Macroglobulinemia | interventions — bazlitoran

ARMS (1):
- IMO-8400 at escalating dose levels (Experimental): IMO-8400 at escalating dose levels by subcutaneous injection
  Interventions: Drug: IMO-8400

INTERVENTIONS:
Drug: IMO-8400 — IMO-8400 at escalating dose levels by subcutaneous injection

SUMMARY:
Recent reports have identified a specific oncogenic mutation L265P of the MYD88 gene in approximately 90% of the patients with Waldenström's macroglobulinemia. MYD88 is a key linker protein in the signaling pathway of Toll Like Receptors (TLRs) 7, 8, and 9, and IMO-8400 is an oligonucleotide specifically designed to inhibit TLRs 7,8, and 9. The scientific hypothesis for use of IMO-8400 to treat patients with Waldenström's macroglobulinemia depends on the inhibition of mutant MYD88 signaling in the TLR pathway, thereby interrupting the proliferation of cell populations responsible for the propagation of the disease.

DETAILED DESCRIPTION:
Eligible subjects will be enrolled and assigned to escalating dose cohorts. Treatment will be administered by subcutaneous injection.

ELIGIBILITY:
Inclusion Criteria:

Patients must have a diagnosis of relapsed Waldenstrom's Macroglobulinemia.

In addition to the above, key inclusion and exclusion criteria are listed below.

Inclusion Criteria:

1. At least 18 years of age.
2. Agree to use contraception
3. Hemoglobin ≥ 7.5 g/dL, - Absolute neutrophil count ≥ 1.0 x 109/L (1000/mm3), - Platelets ≥ 50,000/μL

Exclusion Criteria:

1. Is nursing or pregnant
2. Has BMI > 34.9 kg/m2.
3. Has a positive test for human immunodeficiency virus (HIV-1 or -2) hepatitis C virus (HCV) or hepatitis B surface antigen (HBsAg).
4. Receiving chronic systemic corticosteroid therapy > 20 mg of prednisone daily.
5. Being treated with other anti-cancer therapies (approved or investigational).
6. Has, at the initiation of study drug, received cytotoxic chemotherapy or a Bruton's tyrosine kinase (BTK)-inhibitor (e.g. ibrutinib) within the past 3 weeks or rituximab within the past 2 months
7. Has an active infection requiring systemic antibiotics.
8. Has had surgery requiring general anesthesia within 4 weeks of starting the study.
9. Has autoimmune cytopenia (anemia, thrombocytopenia, leukopenia).
10. Has heart failure of Class III or IV.
11. Has sensory or motor neuropathy limiting daily activities.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2014-03; Primary Completion 2017-04 (Actual); Study Completion 2017-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Cornfeld, MD, MPH, Study Director — Idera Pharmaceuticals, Inc.
Locations (10):
- United States (10):
  - Cancer Centers of Excellence, Fayetteville, Arkansas
  - UCLA, Los Angeles, California
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - Emory Winship Cancer Institute, Atlanta, Georgia
  - Horizon BioAdvance, Lafayette, Indiana
  - Mayo Clinic, Rochester, Minnesota
  - Hackensack University, Hackensack, New Jersey
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - MD Anderson Cancer Center, Houston, Texas
  - Seattle Cancer Care Alliance, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were enrolled from 02 April 2014 through 31 March 2017 at 14 study sites in the United States.
Pre-assignment Details: Screening occurred ≤ 21 days before Day 1 (the first injection of study drug).
Groups:
- IMO-8400 0.6 mg/kg 1x/wk: IMO-8400 0.6 mg/kg once weekly s.c.
- IMO-8400 1.2 mg/kg 1x/wk: IMO-8400 1.2 mg/kg once weekly s.c.
- IMO-8400 1.2 mg/kg 2x/wk: IMO-8400 1.2 mg/kg twice weekly s.c.
- IMO-8400 2.4 mg/kg 1x/wk: IMO-8400 2.4 mg/kg once weekly s.c.
Period: Overall Study
Arm/Group | IMO-8400 0.6 mg/kg 1x/wk | IMO-8400 1.2 mg/kg 1x/wk | IMO-8400 1.2 mg/kg 2x/wk | IMO-8400 2.4 mg/kg 1x/wk
Started | 6 | 5 | 14 | 6
Completed | 5 | 2 | 5 | 0
Not Completed | 1 | 3 | 9 | 6
Not completed — Adverse Event | 0 | 0 | 4 | 2
Not completed — Lack of Efficacy | 0 | 2 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 2 | 1
Not completed — Study terminated by Sponsor | 0 | 0 | 0 | 2
Not completed — Miscellaneous | 1 | 1 | 2 | 1

BASELINE CHARACTERISTICS:
Population: Safety Population
Groups:
- Total: Total of all reporting groups
Arm/Group | IMO-8400 0.6 mg/kg 1x/wk | IMO-8400 1.2 mg/kg 1x/wk | IMO-8400 1.2 mg/kg 2x/wk | IMO-8400 2.4 mg/kg 1x/wk | Total
Number analyzed (Participants) | 6 | 5 | 14 | 6 | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 74.8 (12.92) | 70.4 (9.71) | 66.5 (11.17) | 62.7 (11.36) | 68.0 (11.53)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 3 | 1 | 9
  Male | 4 | 2 | 11 | 5 | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 6 | 5 | 14 | 6 | 31
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 0 | 1
  White | 6 | 5 | 12 | 5 | 28
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 5 | 14 | 6 | 31
Time Since WM Diagnosis (yrs) [Mean (Standard Deviation); unit: years] | 7.03 (4.62) | 10.16 (6.90) | 7.66 (3.55) | 5.78 (5.22) | 7.58 (4.66)
Baseline IPSSWM Score [Count of Participants; unit: Participants]
  Low | 2 | 1 | 5 | 2 | 10
  Intermediate | 3 | 3 | 8 | 4 | 18
  High | 1 | 1 | 1 | 0 | 3
Baseline Total IgM [Mean (Standard Deviation); unit: mg/dL] — Population: Total IgM was not collected in the original protocol version, and only added after a protocol amendment.
  mg/dL
    number analyzed (Participants) | 1 | 5 | 14 | 6 | 26
    (all) | 1090 (NA) — N=1 | 2410 (973) | 2857 (1567) | 2910 (1727) | 2715 (1473)
Baseline Monoclonal IgM [Mean (Standard Deviation); unit: g/dL] | 1.04 (0.640) | 0.93 (0.614) | 1.57 (0.835) | 1.62 (0.741) | 1.37 (0.773)

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability of IMO-8400 in Patients With Waldenstrom's Macroglobulinemia
Description: Safety and tolerability of IMO-8400 in patients with Waldenstrom's Macroglobulinemia: Assessment of adverse events
Time Frame: Up to 24 weeks
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | IMO-8400 0.6 mg/kg 1x/wk | IMO-8400 1.2 mg/kg 1x/wk | IMO-8400 1.2 mg/kg 2x/wk | IMO-8400 2.4 mg/kg 1x/wk
Number analyzed (Participants) | 6 | 5 | 14 | 6
Participants
  At Least 1 TEAE | 6 | 5 | 14 | 6
  At Least 1 Related TEAE | 5 | 2 | 12 | 6
  At Least 1 Grade >=3 TEAE | 1 | 2 | 7 | 3
  At Least 1 SAE | 0 | 0 | 1 | 2
  At Least 1 DLT | 0 | 0 | 1 | 0
  At Least 1 TEAE Leading to Death | 0 | 0 | 0 | 0
  At Least 1 TEAE Leading to Premature Treatment DC | 0 | 0 | 4 | 2

2. Secondary Outcome: Best Overall Response
Description: Best Overall Response using criteria from the VIth International Workshop in Waldenstrom's Macroglobulinemia
Time Frame: Up to 24 weeks
Population: Efficacy Evaluable Population
Measure: Count of Participants; unit: Participants
Arm/Group | IMO-8400 0.6 mg/kg 1x/wk | IMO-8400 1.2 mg/kg 1x/wk | IMO-8400 1.2 mg/kg 2x/wk | IMO-8400 2.4 mg/kg 1x/wk
Number analyzed (Participants) | 5 | 4 | 12 | 5
Participants
  Complete Response | 0 | 0 | 0 | 0
  Very Good Partial Response | 0 | 0 | 0 | 0
  Partial Response | 1 | 0 | 2 | 0
  Minor Response | 2 | 0 | 4 | 1
  Standard Deviation | 2 | 3 | 4 | 3
  Progressive Disease | 0 | 1 | 1 | 1
  Not Evaluable | 0 | 0 | 1 | 0

3. Secondary Outcome: Identify the Number of Patients Experiencing DLTs at Each Dose Level
Description: To identify an appropriate dose of IMO-8400 for further clinical evaluation via evaluation of DLT at each dose level
Time Frame: 28 days
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | IMO-8400 0.6 mg/kg 1x/wk | IMO-8400 1.2 mg/kg 1x/wk | IMO-8400 1.2 mg/kg 2x/wk | IMO-8400 2.4 mg/kg 1x/wk
Number analyzed (Participants) | 6 | 5 | 14 | 6
Participants | 0 | 0 | 1 | 0

4. Secondary Outcome: Pharmacokinetics of Escalating Dose Levels of IMO 8400 Administered by SC Injection - Cmax.
Description: Pharmacokinetics of escalating dose levels of IMO 8400 administered by SC injection - Cmax.
Time Frame: Cycle 1 Week 1 Day 1: Samples were obtained pre-dose (within 1 hr prior to injection) and post-dose at 1 hr (+/-5 min), 2 hrs (+/-10 min) and 4 hrs (+/-15 min)
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Cmax (ng/mL)
Arm/Group | IMO-8400 0.6 mg/kg 1x/wk | IMO-8400 1.2 mg/kg 1x/wk | IMO-8400 1.2 mg/kg 2x/wk | IMO-8400 2.4 mg/kg 1x/wk
Number analyzed (Participants) | 6 | 5 | 14 | 6
Cmax (ng/mL) | 807.6 (70.3) | 2137.9 (68.7) | 2421.2 (50.8) | 4433.1 (29.9)

5. Secondary Outcome: Pharmacokinetics of Escalating Dose Levels of IMO 8400 Administered by SC Injection - AUC0-t (hr*ng/mL)
Description: Pharmacokinetics of escalating dose levels of IMO 8400 administered by SC injection - AUC0-t (hr*ng/mL) .
Time Frame: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: AUC0-t (hr*ng/mL)
Arm/Group | IMO-8400 0.6 mg/kg 1x/wk | IMO-8400 1.2 mg/kg 1x/wk | IMO-8400 1.2 mg/kg 2x/wk | IMO-8400 2.4 mg/kg 1x/wk
Number analyzed (Participants) | 6 | 5 | 14 | 6
AUC0-t (hr*ng/mL) | 2565.8 (64.6) | 6493.0 (61.7) | 7229.3 (54.5) | 13691.7 (32.3)

ADVERSE EVENTS:
Time Frame: From obtaining informed consent through EOS visit. (up to 24 weeks)
Arm/Group | IMO-8400 0.6 mg/kg 1x/wk | IMO-8400 1.2 mg/kg 1x/wk | IMO-8400 1.2 mg/kg 2x/wk | IMO-8400 2.4 mg/kg 1x/wk
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/5 | 0/14 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/5 | 1/14 | 2/6
Other Adverse Events (participants affected / at risk) | 6/6 | 5/5 | 13/14 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IMO-8400 0.6 mg/kg 1x/wk (N=6) | IMO-8400 1.2 mg/kg 1x/wk (N=5) | IMO-8400 1.2 mg/kg 2x/wk (N=14) | IMO-8400 2.4 mg/kg 1x/wk (N=6)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | IMO-8400 0.6 mg/kg 1x/wk (N=6) | IMO-8400 1.2 mg/kg 1x/wk (N=5) | IMO-8400 1.2 mg/kg 2x/wk (N=14) | IMO-8400 2.4 mg/kg 1x/wk (N=6)
Anemia (Blood and lymphatic system disorders) | 0 | 1 | 5 | 0
Lymph node pain (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 2 | 0
Splenomegaly (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
Diplopia (Eye disorders) | 1 | 0 | 0 | 0
Dry eye (Eye disorders) | 0 | 0 | 1 | 1
Eye pruritis (Eye disorders) | 0 | 0 | 1 | 0
Lacrimation increased (Eye disorders) | 0 | 0 | 1 | 0
Vision blurred (Eye disorders) | 0 | 0 | 1 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 2 | 2
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 3 | 3
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Early satiety (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastrointestinal pain (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Impaired gastric emptying (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 1 | 3 | 3
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Chills (General disorders) | 0 | 1 | 2 | 2
Fatigue (General disorders) | 1 | 1 | 5 | 3
Hyperhidrosis (General disorders) | 0 | 0 | 1 | 0
Influenza like illness (General disorders) | 0 | 0 | 1 | 0
Infusion related reaction (General disorders) | 0 | 0 | 2 | 0
Injection site bruising (General disorders) | 0 | 0 | 0 | 1
Injection site erythema (General disorders) | 3 | 0 | 0 | 0
Injection site haemorrhage (General disorders) | 0 | 0 | 0 | 1
Injection site nodule (General disorders) | 0 | 0 | 1 | 0
Injection site pain (General disorders) | 2 | 0 | 1 | 0
Injection site pruritis (General disorders) | 0 | 1 | 0 | 0
Injection site reaction (General disorders) | 1 | 1 | 5 | 4
Malaise (General disorders) | 0 | 0 | 1 | 0
Oedema (General disorders) | 0 | 0 | 1 | 0
Pain (General disorders) | 0 | 0 | 1 | 1
Pyrexia (General disorders) | 0 | 1 | 1 | 3
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Hypogammaglobulinaemia (Infections and infestations) | 0 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 0
Cystitis (Infections and infestations) | 0 | 0 | 0 | 1
Lung Infection (Infections and infestations) | 0 | 0 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 3 | 2
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 1 | 0 | 0 | 0
Cardiac murmur (Investigations) | 1 | 0 | 0 | 0
Hepatic enzyme increased (Investigations) | 0 | 0 | 1 | 0
Inspiratory capacity decreased (Investigations) | 0 | 0 | 0 | 1
Intraocular pressure test abnormal (Investigations) | 1 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 1 | 0
Platelet count decreased (Investigations) | 0 | 0 | 1 | 0
Spinal myelogram (Investigations) | 0 | 0 | 0 | 1
Weight decreased (Investigations) | 1 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 2 | 2
Dehydration (Metabolism and nutrition disorders) | 2 | 0 | 1 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 3
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 3
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Gout (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1 | 3
Brachial plexopathy (Nervous system disorders) | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 2 | 2
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 2 | 3 | 2
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 1
Memory impairment (Nervous system disorders) | 0 | 0 | 1 | 0
Neuralgia (Nervous system disorders) | 0 | 0 | 1 | 1
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 1 | 1
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0 | 2 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 1
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 1 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 2
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 0 | 0
Haematoma (Vascular disorders) | 1 | 0 | 2 | 1
Hot flush (Vascular disorders) | 0 | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Idera staff in collaboration with the Investigator will be responsible for writing presentations and manuscripts for publication. Investigators will not be allowed to publish or present the data from this study without prior agreement with Idera.

DOCUMENTS (2):
  • Study Protocol (2016-03-14): https://cdn.clinicaltrials.gov/large-docs/09/NCT02092909/Prot_000.pdf
  • Statistical Analysis Plan (2017-04-21): https://cdn.clinicaltrials.gov/large-docs/09/NCT02092909/SAP_001.pdf